CLINICAL TRIAL: NCT04586166
Title: SASS: Randomized Trial of Single-incision Versus Retropubic Mid-Urethral Sling (Solyx) for Concomitant Management of Stress Urinary Incontinence During Minimally Invasive Sacrocolpopexy
Brief Title: Single-incision Versus Retropubic Mid-Urethral Sling (Solyx) for SUI During Minimally Invasive Sacrocolpopexy
Acronym: SASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00068839
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor Disorders
Keywords: Retropubic Sling; Single-Incision Sling; Sacrocolpopexy
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked during the five-year follow-up period. Precautions will be taken to minimize unmasking the study groups. Since RP (retropubic) slings require two suprapubic stab incisions, identical sham incision will also be performed in the SIS (Single-Incision Sling) group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RP Sling Group (Experimental): Participants assigned to the retropubic (RP) sling group will have the RP sling placement procedure
  Interventions: Device: RP Sling
- SIS Group (Experimental): Participants assigned to the single-incision sling (SIS) group will have the SIS placement procedure
  Interventions: Device: SIS

INTERVENTIONS:
Device: RP Sling — Participants assigned to the retropubic (RP) sling group will have the RP sling placement procedure.
  Other Names: Advantage RP Sling
  Arms: RP Sling Group
Device: SIS — Participants assigned to the single-incision sling (SIS) group will have the SIS placement procedure.
  Other Names: Solyx SIS System
  Arms: SIS Group

SUMMARY:
SASS (Single-incision Versus Retropubic Mid-Urethral Sling (Solyx) for SUI During Minimally Invasive Sacrocolpopexy) will be a multicenter, prospective, randomized, single-blind non-inferiority trial.

DETAILED DESCRIPTION:
SASS aims to compare the efficacy of a single-incision (SIS) versus a retropubic mid-urethral sling (RP) placed at the time of minimally invasive sacrocolpopexy in women with pelvic organ prolapse and objectively confirmed stress urinary incontinence (SUI).

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Vaginal bulge symptoms as indicated by an affirmative response of >1 to question 3 of the PFDI-SF20
* POP ≥ stage II according to the pelvic organ prolapse quantification (POP-Q) system45, with evidence of apical descent
* Women being considered for minimally invasive sacrocolpopexy (with or without concomitant hysterectomy)
* Objective SUI: positive standardized cough stress test on clinical examination or on urodynamic study with reduced prolapse
* Understanding and acceptance of the need to return for all scheduled follow-up visits and willing to complete study questionnaires
* Able to give informed consent

Exclusion Criteria:

* Prior surgery for stress urinary incontinence including mid-urethral sling; Burch/MMK; fascial pubovaginal sling (autologous, xenograft or allograft); and urethral bulking injection
* Any serious disease, or chronic condition, that could interfere with the study compliance
* Unwilling to have a synthetic sling
* Untreated and unresolved urinary tract infection
* Poorly-controlled diabetes mellitus (HgbA1c > 9 within 3 months of surgery date)
* Neurogenic bladder/ pre-operative self-catheterization
* Elevated post-void residual/PVR (>150 ml) that does not resolve with prolapse reduction testing (pessary, prolapse reduced uroflow or micturition study)
* Prior pelvic radiation
* Inflammatory bowel disease
* Current genitourinary fistula or urethral diverticulum
* Planned concomitant bowel related surgery including sphincteroplasty and perineal rectal prolapse surgery, rectovaginal fistula repair, hemorrhoidectomy
* Pregnant or Planning to Conceive
* Incarcerated

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with pelvic organ prolapse.
Enrollment: 180 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with subjectively bothersome stress incontinence | 6 weeks after surgery
  Measured by a positive response of > 1 to Question 17 on Pelvic Floor Distress Inventory short form-20 (PFDI-20). Response scale from 0 to 4. Symptoms Not Present = NO 0 = not present Symptoms Present = YES, scale of bother: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit
Number of participants with subjectively bothersome stress incontinence | 1 year after surgery
  Measured by a positive response of > 1 to Question 17 on Pelvic Floor Distress Inventory short form-20 (PFDI-20). Response scale from 0 to 4. Symptoms Not Present = NO 0 = not present Symptoms Present = YES, scale of bother: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit
Number of participants with subjectively bothersome stress incontinence | 3 years after surgery
  Measured by a positive response of > 1 to Question 17 on Pelvic Floor Distress Inventory short form-20 (PFDI-20). Response scale from 0 to 4. Symptoms Not Present = NO 0 = not present Symptoms Present = YES, scale of bother: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit
Number of participants with subjectively bothersome stress incontinence | 5 years after surgery
  Measured by a positive response of > 1 to Question 17 on Pelvic Floor Distress Inventory short form-20 (PFDI-20). Response scale from 0 to 4. Symptoms Not Present = NO 0 = not present Symptoms Present = YES, scale of bother: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale Surgeon ease of Use) | Baseline, Surgery, Post Op: week 2, week 6, year 1, year 2, year 3, and year 5
  This will be assessed using the numeric rating scale (NRS). The score is 0-10, with higher scores denoting a greater degree of satisfaction.
Pelvic Organ Prolapse/Urinary Incontinence Sexual Functioning Short Form (PISQ-IR) | Baseline, Surgery, Post Op: week 2, week 6, year 1, year 2, year 3, and year 5
  Questionnaire consists of 20 questions regarding sexual functioning. PISQ-IR consists of two parts. Part 1, for not Sexually Active (NSA) women, and par 2 for SA women. Response value varies from 1 to 5. Part 1, for not SA (NSA) women, where higher scores indicate a greater impact of the condition on sexual inactivity. Part 2, for SA women, with higher scores indicating better sexual function.
Pelvic Floor Impact (PFIQ-SF7) | Baseline, Surgery, Post Op: week 2, week 6, year 1, year 2, year 3, and year 5
  Consists of 3 scales with each 7 questions and will be used to assess quality of life regarding pelvic floor related quality of life. The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother
Patient Global Impression of Improvement (PGI-I) | Baseline, Surgery, Post Op: week 2, week 6, year 1, year 2, year 3, and year 5
  7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative baseline - lower scores denote improvement - 1= Very much better to 7 = Very much worse
Assessment of post-void residual (PVR) volume | Baseline, Surgery, Post Op: week 2, week 6, year 1, year 2, year 3, and year 5
  Post Void Residual/PVR measurement - (collected via bladder scan or CIC) (Clean Intermittent Catheterization). PVR can be as minimum as 0ml of an average bladder capacity of 400ml
Number of Participants needing Retreatment | 6 month up to 5 year post-surgery
  Surgical intervention for urinary retention (sling lysis) at any time point after surgery
Number of Participants needing bladder drainage | beyond 6 weeks post-surgery
  Requirement of urinary catheter due to incontinence or retention
Pelvic Floor Distress Inventory (PFDI-SF20) | Baseline, Surgery, Post Op: week 2, week 6, year 1, year 2, year 3, and year 5
  The PFDI-20 has a total of 20 questions and 3 scales (Urinary Distress Inventory, Pelvic Organ Prolapse Distress Inventory, and Colorectal-Anal Distress Inventory). The outcomes of this questionnaire will be evaluated stratified by compartment. Each item produces a response of 0 to 4, the average response in each scale is multiplied by 25 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (7):
- United States (6):
  - Florida Robotic and Minimally Invasive Urogynecology, Coconut Creek, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Boston Urogynecology Associates, Cambridge, Massachusetts
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
- Pelvic Floor Foundation of South Africa, University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No
Only limited dataset without PHI will be shared with the study bio statistical group.

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839